CLINICAL TRIAL: NCT01511926
Title: European Study in Patients With Osteoarthritis, Rheumatoid Arthritis, or Ankylosing Spondylitis at Gastrointestinal Risk: A Retrospective, Non-interventional Study of Vimovo™ Prescribing Patterns
Brief Title: Descriptive Study in Patients Treated With Vimovo™, Including Registration of the Physicians' Prescribing Patterns
Acronym: CHARACTERIZE
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D1120C00044
Record Dates: First submitted 2012-01-10; First posted 2012-01-19 (Estimated); Last update posted 2015-03-10 (Estimated); Status verified 2015-03

CONDITIONS: Osteoarthritis; Rheumatoid Arthritis; Ankylosing Spondylitis
Keywords: Vimovo™ treated patients and prescribing patterns; Risk of gastrointestinal side effects
MeSH Terms: conditions — Osteoarthritis; Arthritis, Rheumatoid; Spondylitis, Ankylosing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Adult patients treated with Vimovo™ for diagnosed osteoarthritis (OA), rheumatoid arthritis (RA) or ankylosing spondylitis

SUMMARY:
The most common pain-relievers used by patients with rheumatic disorders are called non-steroidal anti-inflammatory drugs (NSAIDs). These drugs are effective and well documented, but they can cause ulcers and gastrointestinal side effects. Vimovo™ is a tablet containing naproxen (NSAID) and a gastroprotective agent called esomeprazole. Patients with rheumatic disorders, who are at risk for developing gastrointestinal side effects, and where lower doses of naproxen or other NSAID treatment is not considered sufficient, could use this tablet. The regulatory authorities in many European countries have approved the use of Vimovo™, but they would like to understand how various factors influence the doctors' decision to prescribe the tablet and what is characterizing the patients receiving it. The aim of the study is to answer these questions.

DETAILED DESCRIPTION:
European study in patients with osteoarthritis, rheumatoid arthritis, or ankylosing spondylitis at gastrointestinal risk: A retrospective, non-interventional study of Vimovo™ prescribing patterns

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of arthritic disorder (osteoarthritis, rheumatoid arthritis or ankylosing spondylitis) Risk for developing gastrointestinal ulcer Already prescribed Vimovo

Exclusion Criteria:

* Participation in any interventional drug study at the time Vimovo™ was prescribed
* Patients started on Vimovo during the first 3 months after country-specific launch date
* Patients started on Vimovo after the study site is initiated (in order to avoid influence on prescribing decision and recruitment)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients treated with Vimovo™ for diagnosed osteoarthritis (OA), rheumatoid arthritis (RA) or ankylosing spondylitis (AS), and with gastrointestinal (GI) risk factors. The patients will be asked to participate by their treating doctors at GP centres, specialist centres or hospitals across Europe.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2012-01; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Physicians' part of questionnaire score covering speciality, practice setting and NSAIDs prescribing preferences | baseline
Patients' part of questionnaire score covering demography, medical history and Vimovo™ prescribing preferences | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Javier Nuevo, MSC, Study Director — Medical Department, AstraZeneca Spain
Locations (96):
- Belgium (19):
  - Research Site, Aalst
  - Research Site, Dilbeek
  - Research Site, Erembodegem
  - Research Site, Genk
  - Research Site, Halen
  - Research Site, Heers
  - Research Site, Huy
  - Research Site, Langemark
  - Research Site, Lasne
  - Research Site, Lembeke
  - Research Site, Melsele
  - Research Site, Morkhoven
  - Research Site, Olen
  - Research Site, Sart-lez-Spa
  - Research Site, Sint-Lievens-Houtem
  - Research Site, Tessenderlo
  - Research Site, Wambeek
  - Research Site, Wingene
  - Research Site, Zonhoven
- Finland (3):
  - Research Site, Helsinki
  - Research Site, Hyvinkää
  - Research Site, Vantaa
- Germany (10):
  - Research Site, Bad Brückenau
  - Research Site, Blankenhain
  - Research Site, Deggingen
  - Research Site, Freiberg
  - Research Site, Gersthofen
  - Research Site, Hagen
  - Research Site, Lienen
  - Research Site, Löhne
  - Research Site, München
  - Research Site, Stockach
- Netherlands (13):
  - Research Site, 's-Hertogenbosch
  - Research Site, Andijk
  - Research Site, Beek en Donk
  - Research Site, Dordrecht
  - Research Site, Eersel
  - Research Site, Heesch
  - Research Site, Hoogwoud
  - Research Site, Midwoud
  - Research Site, Nijverdal
  - Research Site, Ravenstein
  - Research Site, Sint Geertruid
  - Research Site, Spijkernisse
  - Research Site, Vlodrop
- Norway (14):
  - Research Site, Bøverbru
  - Research Site, Eidsvoll
  - Research Site, Kirkenær
  - Research Site, Kråkerøy
  - Research Site, Oslo
  - Research Site, Røa
  - Research Site, Skarnes
  - Research Site, Sola
  - Research Site, Stavanger
  - Research Site, Strømmen
  - Research Site, Svelvik
  - Research Site, Tananger
  - Research Site, Tønsberg
  - Research Site, Østerås
- Spain (17):
  - Research Site, Las Bayas, Elche, Elche
  - Research Site, Badalona
  - Research Site, Barcelona
  - Research Site, Benaguasil, Valencia
  - Research Site, Elda, Alicante
  - Research Site, Esplugues de Llobregat
  - Research Site, Merida, Badajoz
  - Research Site, Rianxo, A Coruna
  - Research Site, San Fernando, Cadiz
  - Research Site, Santiago de Compostela
  - Research Site, Seville
  - Research Site, Teruel
  - Research Site, Torrelavega, Cantabria
  - Research Site, Valencia
  - Research Site, Vilanova i la Geltrú
  - Research Site, Xativa, Valencia
  - Research Site, Zaragoza
- Switzerland (11):
  - Research Site, Basel
  - Research Site, Bellinzona
  - Research Site, Chur
  - Research Site, Ebmatingen
  - Research Site, Neftenbach / Dorf Neftenbach
  - Research Site, Paradiso
  - Research Site, Sankt Gallen
  - Research Site, Schiers
  - Research Site, Seuzach Dorf
  - Research Site, St. Erhard
  - Research Site, Zurich
- United Kingdom (9):
  - Research Site, Addingham
  - Research Site, Basildon
  - Research Site, Belfast
  - Research Site, Birmingham
  - Research Site, Chippenham
  - Research Site, Heywood
  - Research Site, Randalstown
  - Research Site, Sheffield
  - Research Site, Warminster

REFERENCES:
- See also: Report Synopsis Redacted — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1726&filename=REPORT_SYNOPSIS_D1120C00044_NIS_Report_Redacted.pdf